CLINICAL TRIAL: NCT02043509
Title: Evaluation of a Tailored Text Message Intervention for Pregnant Smokers (MiQuit): a Pilot Trial
Brief Title: MiQuit Trial: Tailored Text Messages for Pregnant Women
Acronym: MiQuit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 13113; 13/EM/0427 (Other: UK Research Ethics Committee)
Record Dates: First submitted 2014-01-14; First posted 2014-01-23 (Estimated); Results first posted 2019-07-15 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-04

CONDITIONS: Pregnancy; Smoking
Keywords: smoking cessation; pregnancy; cessation support; tailored text messages; self-help; MiQuit
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MiQuit (Experimental): 12 weeks of MiQuit text support plus a standard NHS leaflet giving information and advice on stopping smoking in addition to usual care
  Interventions: Behavioral: MiQuit
- Control (No Intervention): Usual care plus the same standard NHS leaflet giving information and advice on stopping smoking

INTERVENTIONS:
Behavioral: MiQuit — MiQuit is an automated responsive text message support programme lasting 12 weeks which provides tailored smoking cessation support and advice to the participant's mobile phone. This support includes motivational messages, advice about preparing for a quit attempt, how to manage cravings and withdrawal, dealing with trigger situations, information about how smoking affects babies and general encouragement.
  Arms: MiQuit

SUMMARY:
The overall aim of the study is to estimate the likely impact of the MiQuit text message based smoking cessation service for pregnant smokers and to establish robust estimates for the key factors which would be required in order to design a larger definitive trial of this intervention(MiQuit).

These key factors include: the range of recruitment rates in different centres; quit rates amongst participants; feasibility of assessing smoking status of participants in later pregnancy; and the likely effect of MiQuit when women are offered this in National Health Service (NHS) settings.

DETAILED DESCRIPTION:
Epidemiological evidence indicates that smoking during pregnancy increases the risk of many pregnancy related complications and is associated with many adverse postnatal problems. Around 15% of women still smoke throughout their pregnancy; younger women and those from more deprived backgrounds are much more likely to smoke. Behavioural support, available through NHS Stop Smoking Services, is effective but only accessed by a minority of smokers with most trying to quit alone. For this large group, self-help interventions may be an effective alternative.

MiQuit is a 12 week tailored, self-help, text-message intervention developed for pregnant smokers. A pilot study found this was feasible and acceptable for recipients, thus if MiQuit could have such an impact in routine NHS care, its low cost would make it highly cost-effective.

Before MiQuit could be used in routine care, a definitive randomised controlled trial (RCT) would be needed but currently there is insufficient information to justify conducting this.

This pilot trial will investigate whether it is possible to evaluate MiQuit in a multi-centre RCT located within the NHS, using research network resources. This study will recruit 400 pregnant smokers who will be randomly allocated to either MiQuit or control, and will provide estimates for the parameters required for determining the necessary resources for a definitive trial. These include: the range of recruitment rates in different centres; quit rates amongst participants; feasibility of assessing smoking status of trial participants in later pregnancy and ascertainment rates obtained; and the likely effect of MiQuit when women are offered this in NHS settings.

Secondary objectives include; To estimate and model the likely effectiveness and cost effectiveness of MiQuit compared with usual care including a generic smoking cessation information leaflet; To document participants' use of MiQuit interactive features and of NHS cessation support; To assess the effect of MiQuit on social cognitive determinants of quitting smoking and; To explore participant views and experiences of using MiQuit.

The participants will be recruited before 25 weeks gestation when they attend NHS hospital clinics for routine antenatal ultrasound scans. Recruitment will take place in around 12 United Kingdom (UK) centres over a 12 month period. Follow-up will be via telephone at 1 month after randomization and again at week 36 gestation. The follow-up is over a 9 month period. If a participant reports they have stopped smoking, this "quit" will be validated with a exhaled Carbon Monoxide (CO) measurement and/or salivary cotinine measurement.

A small number of semi-structured telephone interviews will be carried out with a selection of participants from the MiQuit arm to explore their views and experience of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant and less than 25 weeks gestation
* Smoking at least 5 cigarettes per day pre-pregnancy
* Smoking at least 1 cigarette on a typical day during pregnancy
* Aged 16 or over
* Agrees to accept information to assist cessation
* Has own or has primary use of a mobile phone
* Familiar with sending and receiving text messages
* Able to understand written English (text messages are in English only) and consent issues explained in English.
* Able to give informed consent

Exclusion Criteria:

•Already enrolled in another text service to assist smoking cessation

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2014-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Coleman, Professor, Study Chair — University of Nottingham
Locations (15):
- United Kingdom (15):
  - Mid Cheshire Hospitals NHS Foundation Trust, Crewe, Cheshire
  - Chesterfield Royal Hospitals NHS Foundation Trust, Chesterfield, Derbyshire
  - Derby Hospitals NHS Foundation Trust, Derby, Derbyshire
  - United Lincolnshire Hospitals NHS Trust, Boston, Lincolnshire
  - United Lincolnshire Hospitals NHS Trust, Lincoln, Lincolnshire
  - Nottingham University Hospitals NHS Trust, City Hospital, Nottingham, Nottinghamshire
  - Nottingham University Hospitals NHS Trust, QMC, Nottingham, Nottinghamshire
  - Sherwood Forest Hospitals NHS Foundation Trust, Sutton in Ashfield, Nottinghamshire
  - University Hospital of North Staffordhsire NHS Trust, Stoke-on-Trent, Staffordshire
  - Birmingham Womens NHS Foundation Trust, Birmingham, W Midlands
  - Sandwell & West Birmingham Hospitals NHS Trust, Birmingham, West Midlands
  - The Dudley Group NHS Foundation Trust, Dudley, West Midlands
  - Heart of England NHS Foundation Trust, Birmingham
  - Central Manchester University Hosptitals NHS Foundation Trust, Manchester
  - University Hospitals North Midlands NHS Trust, Stafford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Naughton F, Prevost AT, Gilbert H, Sutton S. Randomized controlled trial evaluation of a tailored leaflet and SMS text message self-help intervention for pregnant smokers (MiQuit). Nicotine Tob Res. 2012 May;14(5):569-77. doi: 10.1093/ntr/ntr254. Epub 2012 Feb 6. PMID 22311960
- [Derived] Cooper S, Foster K, Naughton F, Leonardi-Bee J, Sutton S, Ussher M, Leighton M, Montgomery A, Parrott S, Coleman T. Pilot study to evaluate a tailored text message intervention for pregnant smokers (MiQuit): study protocol for a randomised controlled trial. Trials. 2015 Jan 27;16:29. doi: 10.1186/s13063-014-0546-4. PMID 25622639

RESULTS

PARTICIPANT FLOW:
Period: Baseline to 1st Follow-up
Arm/Group | MiQuit | Control
Started | 203 | 204
Completed | 138 | 157
Not Completed | 65 | 47
Not completed — Lost to Follow-up | 61 | 47
Not completed — Withdrawal by Subject | 4 | 0
Period: Baseline to 2nd Follow-up
Arm/Group | MiQuit | Control
Started (Note that participants who were lost to 1st follow-up could be present at 2nd follow-up.) | 203 | 204
Completed | 129 | 132
Not Completed | 74 | 72
Not completed — Lost to Follow-up | 67 | 67
Not completed — Withdrawal by Subject | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MiQuit | Control | Total
Number analyzed (Participants) | 203 | 204 | 407
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 12 | 22
  Between 18 and 65 years | 193 | 192 | 385
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.6 (5.7) | 26.4 (5.7) | 26.5 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 203 | 204 | 407
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 203 | 204 | 407

OUTCOME MEASURES:

1. Primary Outcome: Continuous Abstinence From Smoking Reported From 4 Weeks Post-randomisation Until Late Pregnancy, Biochemically Validated at Late Pregnancy.
Description: The primary smoking outcome measure will be the number of participants reporting continuous abstinence from smoking from 4 weeks after randomisation until follow up at the end of pregnancy (approximately 36 weeks gestation), validated by exhaled CO and/or saliva cotinine estimation at approximately 36 weeks gestation.
Time Frame: 36 weeks gestation
Population: All participants were included in analysis. Participants lost to follow up were assumed to be smoking.
Measure: Count of Participants; unit: Participants
Arm/Group | MiQuit | Control
Number analyzed (Participants) | 203 | 204
Participants | 11 | 4
Statistical Analysis 1: Comparison: MiQuit vs Control; Test type: Superiority; Adjusted odds ratio = 2.70, 95% CI 2-sided [0.93 to 9.35] — Odds ratios are model-based (adjusted by site and gestation at randomization). 95% profile confidence intervals are reported

2. Secondary Outcome: Continuous Abstinence From Smoking Reported From 4 Weeks Post-randomisation Until Late Pregnancy, Self-report.
Description: The number of participants reporting continuous abstinence from smoking from 4 weeks after randomisation until follow up at the end of pregnancy (approximately 36 weeks gestation), self-reported.
Time Frame: 36 weeks gestation
Population: All participants were included in analysis. Participants lost to follow up were assumed to be smoking.
Measure: Count of Participants; unit: Participants
Arm/Group | MiQuit | Control
Number analyzed (Participants) | 203 | 204
Participants | 33 | 33
Statistical Analysis 1: Comparison: MiQuit vs Control; Test type: Superiority; Adjusted odds ratio = 1.03, 95% CI 2-sided [0.61 to 1.75] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: 7-day Point Prevalence Abstinence From Smoking Reported at Late Pregnancy, Self-report.
Description: The number of participants reporting 7-day abstinence from smoking at the end of pregnancy (approximately 36 weeks gestation), self-reported.
Time Frame: 36 weeks gestation
Population: All participants were included in analysis. Participants lost to follow up were assumed to be smoking.
Measure: Count of Participants; unit: Participants
Arm/Group | MiQuit | Control
Number analyzed (Participants) | 203 | 204
Participants | 36 | 28
Statistical Analysis 1: Comparison: MiQuit vs Control; Test type: Superiority; Adjusted odds ratio = 1.34, 95% CI 2-sided [0.79 to 2.31] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: 7-day Point Prevalence Abstinence From Smoking Reported at Late Pregnancy, Biochemically Validated.
Description: The number of participants reporting 7-day abstinence from smoking at the end of pregnancy (approximately 36 weeks gestation), validated by exhaled CO and/or saliva cotinine estimation.
Time Frame: 36 weeks gestation
Population: All participants were included in analysis. Participants lost to follow up were assumed to be smoking.
Measure: Count of Participants; unit: Participants
Arm/Group | MiQuit | Control
Number analyzed (Participants) | 203 | 204
Participants | 15 | 9
Statistical Analysis 1: Comparison: MiQuit vs Control; Test type: Superiority; Adjusted odds ratio = 1.67, 95% CI 2-sided [0.72 to 4.03] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: 7-day Point Prevalence Abstinence From Smoking Reported at 4 Weeks Post-randomization, Self-report.
Description: The number of participants reporting 7-day abstinence from smoking at 4 weeks after randomisation, self-reported.
Time Frame: 4 weeks post-randomisation
Population: All participants were included in analysis. Participants lost to follow up were assumed to be smoking.
Measure: Count of Participants; unit: Participants
Arm/Group | MiQuit | Control
Number analyzed (Participants) | 203 | 204
Participants | 15 | 7
Statistical Analysis 1: Comparison: MiQuit vs Control; Test type: Superiority; Adjusted odds ratio = 2.11, 95% CI 2-sided [0.89 to 5.46] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: 7-day Point Prevalence Abstinence From Smoking Reported at Both 4 Weeks Post-randomization and at Late Pregnancy, Self-report.
Description: The number of participants reporting 7-day abstinence from smoking at both 4 weeks after randomisation and at follow up at the end of pregnancy (approximately 36 weeks gestation), self-reported.
Time Frame: 36 weeks gestation
Population: All participants were included in analysis. Participants lost to follow up were assumed to be smoking.
Measure: Count of Participants; unit: Participants
Arm/Group | MiQuit | Control
Number analyzed (Participants) | 203 | 204
Participants | 13 | 4
Statistical Analysis 1: Comparison: MiQuit vs Control; Test type: Superiority; Adjusted odds ratio = 3.16, 95% CI 2-sided [1.14 to 10.69] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: 7-day Point Prevalence Abstinence From Smoking Reported at Both 4 Weeks Post-randomization and at Late Pregnancy, Biochemically Validated at Late Pregnancy.
Description: The number of participants reporting 7-day abstinence from smoking at both 4 weeks after randomisation and at follow up at the end of pregnancy (approximately 36 weeks gestation), validated by exhaled CO and/or saliva cotinine estimation at approximately 36 weeks gestation.
Time Frame: 36 weeks gestation
Population: All participants were included in analysis. Participants lost to follow up were assumed to be smoking.
Measure: Count of Participants; unit: Participants
Arm/Group | MiQuit | Control
Number analyzed (Participants) | 203 | 204
Participants | 8 | 2
Statistical Analysis 1: Comparison: MiQuit vs Control; Test type: Superiority; Adjusted odds ratio = 3.28, 95% CI 2-sided [0.90 to 17.36] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Number of 24 Hour Quit Attempts
Description: Number of short-term, 24 hour quit attempts noted per participant, from baseline until follow up at the end of pregnancy (approximately 36 weeks gestation).
Time Frame: 36 weeks gestation
Population: Outcomes are calculated out of 254 participants with response data at late pregnancy follow up (124 MiQuit, 130 Standard Care).
Measure: Median (Inter-Quartile Range); unit: number of events reported
Arm/Group | MiQuit | Control
Number analyzed (Participants) | 124 | 130
number of events reported | 2 [1 to 3] | 1 [0 to 3]
Statistical Analysis 1: Comparison: MiQuit vs Control; Test type: Superiority; p = 0.118, Mann-Whitney U-test

9. Secondary Outcome: Reported Use of NHS and Other (Non-trial) Cessation Support
Description: Reported use of any NHS cessation support or other (non-trial) cessation support (e.g. non-NHS websites), from baseline until follow up at the end of pregnancy (approximately 36 weeks gestation).
Time Frame: 36 weeks gestation
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | MiQuit | Control
Number analyzed (Participants) | 124 | 130
Participants | 83 | 98

10. Secondary Outcome: Number of Requests to Stop Text Support
Description: The number of participants in the trial arm who discontinued the text support prematurely, from baseline until follow up at the end of pregnancy (approximately 36 weeks gestation).
Time Frame: 36 weeks gestation
Population: All participants allocated to the trial arm were included in analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | MiQuit
Number analyzed (Participants) | 203
Participants | 27

ADVERSE EVENTS:
Arm/Group | MiQuit | Control
Serious Adverse Events (participants affected / at risk) | 0/203 | 0/204
Other Adverse Events (participants affected / at risk) | 0/203 | 0/204

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes